CLINICAL TRIAL: NCT04638777
Title: Repetitive Transcranial Magnetic Stimulation With H-coil in Parkinson's Disease: A Double-blind, Placebo-controlled Study
Brief Title: Repetitive Transcranial Magnetic Stimulation With H-coil in Parkinson's Disease (rTMS-PD)
Acronym: rTMS-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giancarlo Comi (Other)
Responsible Party: Sponsor-Investigator, Giancarlo Comi, MD, Principal Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMS-PD
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real rTMS stimulation over M1 and PFC (Active Comparator)
  Interventions: Device: rTMS with H-coil
- Real rTMS stimulation over M1 and sham rTMS over PFC (Active Comparator)
  Interventions: Device: rTMS with H-coil
- Sham rTMS over M1 and PFC (Sham Comparator)
  Interventions: Device: rTMS with H-coil

INTERVENTIONS:
Device: rTMS with H-coil — Real repetitive transcranial magnetic stimulation with H-coil over M1 and PFC
  Arms: Real rTMS stimulation over M1 and PFC
Device: rTMS with H-coil — Real repetitive transcranial magnetic stimulation with H-coil over M1 and sham repetitive transcranial magnetic stimulation with H-coil over PFC
  Arms: Real rTMS stimulation over M1 and sham rTMS over PFC
Device: rTMS with H-coil — Sham repetitive transcranial magnetic stimulation with H-coil over M1 and PFC
  Arms: Sham rTMS over M1 and PFC

SUMMARY:
Focal repetitive transcranial magnetic stimulation (rTMS) has been applied to improve symptoms in Parkinson disease (PD) with conflicting results. However, the stimulation with H-coil has been shown to stimulate a wider cortical area compared with the standard coils, with preliminary results confirming the potential efficacy of the treatment. In this study the investigators aimed to explore the safety and efficacy of excitatory rTMS with H-coil on PD motor symptoms.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled study, with a 1:1:1 randomization into three groups: group 1 - real rTMS over primary motor cortex and prefrontal cortex (M1-PFC): group 2 - real rTMS over M1 and sham rTMS over PFC; group 3 - sham stimulation over both targets

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≤80 years
* Diagnosis of Parkinson's disease according to UK Brain Bank criteria
* Hoehn and Yahr (HY) scale II-IV
* Stable anti-depressive and anti-parkinsonian therapy for at least two months prior to enrollment
* Subjects who answered all questions in the TMS pre-treatment safety questionnaire in a negative manner.
* Have given written informed consent

Exclusion Criteria:

* Presence of an additional neurological or psychiatric pathology
* Severe personality disorder
* Uncontrolled hypertension.
* History of epilepsy, seizures, febrile convulsions.
* History of epilepsy or seizures in first degree relatives.
* History of head injury or stroke.
* Presence of metal prostheses in the head (except dental fillings).
* Metal implants or known history of any metal particles in the eye, cardiac pacemakers, cochlear implants, use of neurostimulators or medical pumps.
* History of migraine within the past six months.
* History of drug or alcohol abuse.
* Impossibility of adequate communication with the examiner.
* Participation in another clinical study, either concomitant or within the previous 3 months.
* Inability to sign the consent form.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2012-06-08 (Actual); Study Completion 2012-07-02 (Actual)

PRIMARY OUTCOMES:
Change at Unified Parkinson's disease rating scale III over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
  A comprehensive 50 question assessment of both motor and non-motor symptoms associated with Parkinson's
Incidence of Treatment-Emergent adverse events [Safety and Tolerability of rTMS] | End of treatment (1 month after start of the treatment)
  monitoring presence of side effects due to the stimulation

SECONDARY OUTCOMES:
Change at Pegboard test over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at Tapping test over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at Up & Go Test over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at dyskinesia rating scale over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at and at Word Fluency test over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at Digit forward & backward test over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at Beck Depression Inventory scale-II over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)
Change at The Clinical Global Impression - Severity scale ( CGI-S) over time | Baseline evaluation, end of treatment (1 month after start of the treatment) and end of follow-up (2 months after start of the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Comi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: ICF, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: data are available from the corresponding author, upon reasonable request